CLINICAL TRIAL: NCT06639412
Title: Enhancing Non-communicable Disease Prevention and Control
Brief Title: Enhancing Non-communicable Disease Prevention and Control Through Parent-Teachers-Development Agents Network in Ethiopia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahir Dar University (Other)
Responsible Party: Principal Investigator, Yeshalem Mulugeta Demilew, Associate professor, Bahir Dar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 17595/24
Record Dates: First submitted 2024-03-13; First posted 2024-10-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Network, Kinship
Keywords: non-communicable diseases; primary health care; Parent-Teachers-Development Agents network
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: A cluster randomized controlled community trial design will also be used to evaluate the effect of Parent-Teachers-Development Agents network.
Who Masked: Outcomes Assessor
Masking Description: outcome assessors will not informed about the intervention and the group to which the intervention is assigned to avoid social desirability bias
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arms (Experimental): The intervention arm will receive the intervention.The intervention will be networking the indigenous parent-teacher association and agriculture development agents with the PHC unit to enhance NCD prevention & control services.
  Interventions: Behavioral: Networking the indigenous parent-teacher association and agriculture development agents with the PHC unit to enhance NCD prevention & control services.
- Control arm (Active Comparator): Control Arm is an arm to which the intervention will not be implemented. The community in the control arm will receive NCD prevention and control measures given through the health care system.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Networking the indigenous parent-teacher association and agriculture development agents with the PHC unit to enhance NCD prevention & control services. — The intervention will be networking the indigenous parent-teacher association and agriculture development agents with the PHC unit to enhance NCD prevention & control services. In this major activity, the project team will establish the network by incorporating agricultural development agents and parents- teacher associations to the health post as foundational actors for educating the community on NCD prevention and control measures. We will implement tier system training to effectively create awareness on NCD and to enhance the NCD care-seeking behavior of the community.
  Arms: Intervention arms
Other: Usual care — The community in the control group will get noncommunicable disease prevention and control measures given through the health care system.
  Arms: Control arm

SUMMARY:
Background: Primary health care is an inclusive, equitable, cost-effective, and efficient approach to enhance the health of the community. Ethiopia has been implementing the primary healthcare approach for the last four decades. However, the performance of primary health care services in the country is not reaching the expected level, mainly in preventing non-communicable diseases.

Objective: The aim of this study is to improve the performance of the primary healthcare system with a focus on preventing non-communicable diseases through the integrated efforts of parent-teachers association and agricultural extension workers with the health extension workers in West Gojjam Zone.

Methods: A cluster randomized controlled community trial and a concurrent cross-sectional quantitative and qualitative approach will be used in this study. The study will be conducted in the West Gojjam Zone among 757 adults. A multistage sampling technique will be used. The intervention will be networking the indigenous parent-teacher association and agriculture development agents with the primary healthcare unit for enhancing non-communicable diseases prevention and control services. A structured interviewer-administered questionnaire will be used to collect quantitative data. Focus group discussions and key informant interviews will be conducted to collect qualitative data. Binary logistic regression analysis and Generalized Estimating Equation with a binary logit function will be computed. Thematic analysis will be used to analyze qualitative data.

Work plan and budget: The project will be conducted from February 2023 to May 2024 using a total 10,000 US dollar.

Benefits and beneficiaries: It will generate evidence on the contribution of networking institutions, community members, and the healthcare system to prevent and lower the burdens of major non-communicable diseases. Ministry of Health, Regional Health Bureaus, Zonal Health Departments, Woreda Health Offices, primary health care units, partners, and stockholders are potential beneficiaries of the project outputs.

DETAILED DESCRIPTION:
Background and rationale Primary Health Care is a whole-of-society approach to health that aims at ensuring the highest possible level of health and well-being and their equitable distribution by focusing on people's needs and as early as possible along the continuum from health promotion and disease prevention to treatment, rehabilitation, and palliative care, and as close as feasible to people's everyday environment (1). Primary Health care (PHC) is a path towards achieving universal health coverage (UHC), health-related sustainable development goals (SDGs), and health security (2). Enhancing PHC interventions across low and middle-income countries could save 60 million lives and increase average life expectancy by 3.7 years by 2030 (1).

Ethiopia has been implementing the PHC approach since the mid-1970s. The three interrelated and synergistic components of PHC are comprehensive integrated health services, multi-sectorial policies, and empowering communities for increased social participation (2). Though there have been noticeable changes in PHC services coverage in Ethiopia, the UHC Index remains at 43% (3).

Ethiopia is in both demographic & epidemiologic shifts with the burden of non-communicable diseases (NCDs) is steadily increasing & is expected to grow at an alarming rate in the next couple of decades (4). In Ethiopia, the prevalence of NCDs ranges from 19-35%. The pooled prevalence of Diabetes Mellitus is 5%, cardiovascular conditions ranged from 13.4 to 32.2%, cancer mortality ranged from 4 to 18%, and respiratory conditions ranged from 1-18% (4).

Non-communicable diseases are lifelong chronic diseases that result in huge morbidity & mortality as well as catastrophic health care cost. Nearly half of all deaths in Ethiopia are attributable to NCDs & injuries. Ethiopian citizens have 18.3% risk of dying prematurely from one of the four main NCDs. The economic loss due to NCDs is 31.3 billion birr annually (5). Hence, NCDs are very serious problems resulting in high burdens to patients, families, communities, and the country at large (4).

The risk factors of NCDs are unhealthy dietary habits, sedentary lifestyle, risky sexual behavior, tobacco use, drinking alcohol, and Khat chewing (5). Low community awareness about NCDs, poor trend of early screening for NCDs, and low NCD service-seeking practices are key challenges contributing to the high prevalence & complications of NCDs. Moreover, most of the cases are unaware of their conditions and come to health care services after the advanced stage (5). This problem is worst in rural communities.

Non-communicable diseases prevention & control is one of the nine essential healthcare packages in the Ethiopian primary healthcare system taking the high burden of NCDs & their serious consequences into consideration (6). Even though NCD care has gotten attention at the policy level in recent years, there are a lot of gaps in implementing NCD prevention & treatment services at the PHC level (7). Evidence show the importance of bringing non-health sectors on board for the national NCD response (7).

Therefore, this study will provide community-wide education aiming to promote healthy living & increasing NCDs care-seeking behavior of the community through training the indigenous administrative & societal structures & networking them with existing PHC units. Parent-Teachers-Development Agents network will be established using the existing social structures. Parent Teachers association from the community and education sector, developmental agents (DAs) from the agriculture sector, health extension workers from the primary healthcare unit, and health development Army from the community. All of them usually reside at the same camp or village and networking these structures is a feasible and cost-effective strategy to implement NCDs prevention and control strategies since multisectoral collaboration is the backbone of PHC service.

Objectives: To determine non-communicable disease care-seeking behavior of the community in West Gojjam Zone, Ethiopia, 2023 To assess knowledge of the community on non-communicable diseases prevention and control measures in West Gojjam Zone, Ethiopia, 2023 To explore barriers interfering non-communicable diseases care-seeking behavior of the community in West Gojjam Zone, Ethiopia, 2023 To establish and implement a Parent-Teachers-Development Agents network to enhance NCDs prevention and control in West Gojjam Zone, Ethiopia, 2023 To evaluate the effectiveness of Parent-Teachers-Development Agents network on non-communicable diseases prevention and control in West Gojjam Zone, Ethiopia, 2023 Scope of the project: Both quantitative and qualitative data will be collected to generate evidence on knowledge, health-seeking behavior, barriers, and effectiveness of the Parent-Teachers-Development Agents networking in preventing and controlling NCDs in West Gojjam Zone.

Beneficiaries of the project: The community, Ministry of Health, Regional Health Bureaus, Zonal Health Departments, Woreda Health Offices, PHCUs, and partners are potential beneficiaries of the project outputs.

Deliverables: The Bahir Dar University team will deliver the following assignments during the consultancy period:

* Develop NCD intervention guideline for the networking on NCDs prevention and control
* Establish the Parent-Teachers-Development Agents network
* Submit inception report about field activities such as data collection, data quality activities, implementation of the intervention and measures taken to challenges faced during implementation to the IPHC-E
* Submit the final report to the IPHC-E
* Submit four manuscripts to a peer-reviewed journal involving the IPHC staff
* Submit a one-page issue brief to the IPHC-E Methods and materials The study will be conducted in the West Gojjam Zone, Amhara Region from February 2023 to May 2024. This study will apply a mixed study design. A concurrent cross-sectional quantitative & qualitative approach will apply to assess the knowledge & NCD care-seeking behavior of the community. Community NCD care-seeking behavior will be assessed using the socioecological model as a guiding framework. A cluster randomized controlled community trial design will also be used to evaluate the effect of Parent-Teachers-Development Agents network.

All adult community members in the West Gojjam zone will be the source population whereas the study population will be all adults over 18 years old in selected Kebeles (the smallest administrative units in Ethiopia). Adults who live at least 6 months in selected Kebeles will be included in the study. A qualitative study will be conducted among purposively selected residents, health care providers, and NCD focal persons. A sample size of 757 is determined using single population proportion formula to determine knowledge & health-seeking behavior (8). G power software is used to determine the sample size for the intervention and 253 participants in the intervention group and 253 respondents in the control group will participate (8).

A multistage sampling technique will be used to determine knowledge & health seeking behavior while a cluster sampling technique will be employed for the intervention. An equal number of clusters (Kebeles) will be allocated into intervention &control clusters using simple randomization &one-to-one ratio (intervention and control arms). A structured interviewer-administered questionnaire will be used to collect quantitative data using Open Data Kit. Focus group discussions among community members & key informant interviews among health professionals & NCD focal persons will be conducted until information saturation using interview guides. Endline data will be collected after three months of intervention implementation.

The intervention will be networking the indigenous parent-teacher association and agriculture development agents with the PHC unit to enhance NCD prevention & control services. In this major activity, the project team will establish the network by incorporating agricultural development agents and parents- teacher associations to the health post as foundational actors for educating the community on NCD prevention and control measures. We will implement tier system training to effectively create awareness on NCD and to enhance the NCD care-seeking behavior of the community.

After establishing the network, first, the research team will provide five days training for the network members using a training guide, role-play, & fieldwork practices. Trained network members will educate the community using indigenous social networks like churches, equb, edir, and senbetie. They will educate the community using education guide, which is prepared in the local language. Leaflets, broachers, & billboards regarding NCD prevention & control measures will be prepared & used. Second, trained teachers will train students on NCD prevention & control measures then students will disseminate the information to their families and neighbors. Third, agricultural workers will educate the community about the importance of the production & consumption of fruits and vegetables as well as food safety measures in the prevention of NCDs. Health extension workers and health development Army will closely supervise the implementation of intervention. Community engagement using existing social structures may require to prevent NCDs.

The intervention will be implemented for 30 minutes every week for three months. The community in the control group will receive routine health care given through the health system. Fidelity checks and other quality assurance measures will be implemented before, during, & after the implementation of the project. The expected outcomes of this intervention will be improved knowledge and NCD care-seeking behavior of the community. Descriptive statistics will be done using SPSS. Binary logistic regression analysis will be used to assess factors associated with knowledge and NCD care-seeking behavior of the community. Generalized Estimating Equation with a binary logit function will be also computed to examine the intervention effects. Thematic analysis will be used to analyze qualitative data. The Institutional Review Board of Bahir Dar University will approve this study.

ELIGIBILITY:
Inclusion Criteria:

-All adult individuals residing in the kebele will be included in the study.

Exclusion Criteria:

-none

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
NCD care-seeking behavior of the community ( number of individuals who screened for NCD) | nine months
  NCD seeking service utilization of the community (checking blood pressure, blood glucose level, cervical cancer screening)
knowledge on NCD | nine months
  improved knowledge of the community about NCD will be assessed using knowledge assessment questions.

SECONDARY OUTCOMES:
Hypertension | nine months
  Reduced blood pressure level

CONTACTS AND LOCATIONS:
Overall Officials: Getu D Alene, PhD, Study Director — Bahir Dar University
Locations (1):
- Bahir Dar University, Bahir Dar, Ethiopia

REFERENCES:
- [Derived] Demilew YM, Wassie GT, Guadie HA, Asemahagn MA, Anagaw TF, Alene GD, Kassie GM. The effect of health education on hypertension, diabetes mellitus, and cervical cancer screening service utilization among eligible adults in a district around Bahir Dar city, Ethiopia: a cluster randomized controlled community trial. BMC Public Health. 2025 Aug 12;25(1):2736. doi: 10.1186/s12889-025-23841-7. PMID 40797194
- See also: Assefa Y, Hill PS, Gilks CF, Admassu M, Tesfaye D, Damme WV. Primary health care contributions to universal health coverage, Ethiopia. Bull World Health Organ. 2020;98:doi: http://dx.doi.org/10.2471/BLT.19.248328:894-905A — http://dx.doi.org/10.2471/BLT.19.248328
- See also: Tesfay FH, Zorbas C, Alston L, Backholer K, Bowe SJ, Bennett CM. Prevalence of chronic non-communicable diseases in Ethiopia: A systematic review and meta-analysis of evidence. Front Public Health. 2022;10:936482.doi: 10.3389/fpubh.2022. — https://doi.org/10.3389/fpubh.2022.936482